CLINICAL TRIAL: NCT06033742
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of HS-10374 in Healthy Subjects
Brief Title: A First in Human Study to Evaluate Safety, Tolerability, Pharmacology of HS-10374 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: HS-10374-101
Record Dates: First submitted 2023-08-24; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-08

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HS-10374 (Experimental): Single and multiple ascending doses of HS-10374 orally
  Interventions: Drug: HS-10374 tablets
- Placebo (Placebo Comparator): Single and multiple ascending doses of HS-10374-matched placebo orally
  Interventions: Drug: HS-10374-matched placebo tablets

INTERVENTIONS:
Drug: HS-10374 tablets — Single or multiple dosing of HS-10374 orally in a fasting state
  Arms: HS-10374
Drug: HS-10374-matched placebo tablets — Single or multiple dosing of HS-10374-matched placebo orally in a fasting state
  Arms: Placebo

SUMMARY:
The purpose of this first-in-human study is to evaluate the safety, tolerability, and pharmacokinetics (PK) of HS-10374 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female subjects between the ages of 18-45 years
2. Have no reproductive potential; or agree to use a highly effective method of contraception, and refrain from donating sperm or eggs during the study period and for at least 6 months after last dosing
3. Have signed the informed consent form approved by the IRB

Exclusion Criteria:

1. Have a clinically significant infection currently or within past 30 days, or have a history of active tuberculosis; or have positive screening test for infectious disease, including tuberculosis, viral hepatitis, AIDS and syphilis
2. Have a history of or current allergic disease
3. Have a history of drug or alcohol abuse or currently positive test result(s) for alcohol or drugs of abuse
4. Smokers smoked ≥5 cigarettes per day within past 3 months or have a positive test result for nicotine
5. Clinically significant abnormal physical examination, vital signs, clinical laboratory values, ECGs or imaging tests
6. Pregnant or breastfeeding female subjects
7. Have received hormone-based contraceptives, drugs that prolong the QT interval, drugs that may cause drug interactions with investigational product, immunosuppressants, vaccines or other drugs within a specific period

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2021-11-13 (Actual); Primary Completion 2023-03-24 (Actual); Study Completion 2023-03-24 (Actual)

PRIMARY OUTCOMES:
Incidence, severity and association with the study drug of adverse events (AEs), serious AEs (SAEs), and AEs leading to discontinuation | Day 1 up to Day 12 (SAD), Day 1 up to Day 42 (MAD)
Number of participants with clinical laboratory abnormalities | Day 1 up to Day 12 (SAD), Day 1 up to Day 42 (MAD)
  Clinical laboratory tests include hematology, urinalysis, stool analysis, blood chemistry, coagulation testing, Cystatin C, urine β2-microglobulin, erythrocyte sedimentation rate, C-reactive protein, etc.
Number of participants with abnormalities of vital signs | Day 1 up to Day 12 (SAD), Day 1 up to Day 42 (MAD)
  Vital sign measured include blood pressure, pulse rate, temperature, and respiration rate.
Number of participants with abnormalities of physical examination | Day 1 up to Day 12 (SAD), Day 1 up to Day 42 (MAD)
  Physical examination includes assessments of general appearance, skin, lymph nodes, head, neck, lung, heart, abdomen, spine, extremities, nervous system, etc.
Number of participants with abnormalities of electrocardiogram (ECG) parameters | Day 1 up to Day 12 (SAD), Day 1 up to Day 42 (MAD)
  ECG parameters include heart rate, PR interval, RR interval, QRS duration, QTcF interval.

SECONDARY OUTCOMES:
Cmax | Day 1 up to Day 6 (SAD), Day 1 up to Day 19 (MAD)
  Maximum plasma concentration
Tmax | Day 1 up to Day 6 (SAD), Day 1 up to Day 19 (MAD)
  Time to reach Cmax
AUC | Day 1 up to Day 6 (SAD), Day 1 up to Day 19 (MAD)
  Area under the plasma concentration-time curve
t½ | Day 1 up to Day 6 (SAD), Day 1 up to Day 19 (MAD)
  Terminal half-life
CL/F | Day 1 up to Day 6 (SAD), Day 1 up to Day 19 (MAD)
  Apparent clearance
Vz/F | Day 1 up to Day 6 (SAD), Day 1 up to Day 19 (MAD)
  Apparent volume of distribution
Rac | Day 1 up to Day 6 (SAD), Day 1 up to Day 19 (MAD)
  Accumulation ratio

CONTACTS AND LOCATIONS:
Overall Officials: Jing Zhang, PhD, Principal Investigator — Huashan Hospital; Jinhua Xu, MD, Principal Investigator — Huashan Hospital
Locations (1):
- Huashan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality, China